CLINICAL TRIAL: NCT04223557
Title: Non-invasive Focused Power Ultrasound Mediated Inferior Perirenal Fat Ablation for Lowering Serum Cholesterol
Brief Title: A Cholesterol Lowering Therapy of Focused Power Ultrasound Mediated Perirenal Fat Ablation
Acronym: CONCISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiangqing Kong, Head of Cardiology,Director,Clinical Professor,Principal Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-SR-388
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Visceral Obesity; Ultrasound Therapy; Dyslipidemias
Keywords: Perirenal fat; Ultrasound Therapy; Dyslipidemias; low-density lipoprotein cholesterol
MeSH Terms: conditions — Obesity, Abdominal; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, sham-controlled study.The ratio of the treatment group versus sham-control group was 2:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FPU treatment (Experimental): Transcutaneous non-invasive ultrasound will be administered to the peri-renal fat for one time via a focused power ultrasound system (FPU) device.
  Interventions: Device: focused power ultrasound treatment
- Sham treatment (Sham Comparator): Partcipates will receive the same procedure as those in experimental arm except that the device will not be activated.
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: focused power ultrasound treatment — Patients will be placed in the lateral decubitus position and receive treatment with sequential bilateral PRF ablation. Before the treatment, a professional sonographer will be responsible for the length, thickness, and width of PRF sac measurement and localisation, and utilise the ultrasonic diagnostic transducer to delineate the targeted region. The treatment will launch layer-by-layer. After confirming accurate localization of the treatment, layer-by-layer PRF ablation will be performed on the patients. The device generates and delivers a pattern of conic-shaped ultrasound energy to the PRF sac noninvasively. The treatment of FPU-mediated PRF ablation will be implemented once.
  Arms: FPU treatment
Device: Sham treatment — Participants will receive the same procedure as those in the FPU treatment including PRF ultrasonic measurement and localization and focused ultrasound treatment parameters setting, except that no energy will be delivered to the PRF.
  Arms: Sham treatment

SUMMARY:
The goal of this clinical trial is to learn about focused power ultrasound (FPU)-mediated perirenal fat (PRF) ablation for lowering serum cholesterol levels. The main questions it aims to answer are:

What is the efficacy, safety, and tolerability of focused power ultrasound (FPU)-mediated perirenal fat ablation for lowering low-density lipoprotein cholesterol (LDL-C) levels? Participants will randomly receive PRF ablation or sham treatment, and undergo follow-up at 24 hours, 1 month, and 3 months post-procedure.

DETAILED DESCRIPTION:
This study aims to evaluate and validate the efficacy and safety of the therapeutic approach of PRF ablation-executed by an externally delivered, completely non-invasive FPU-on serum cholesterol levels in patients with dyslipidaemia, with a low-to-moderate 10-year overall risk of ASCVD.

This is an investigator-initiated, single site, randomised, double-blinded, sham-controlled clinical trial. Further eligibility assessment will be performed at the secondary screening, which has the same design as the baseline examination. Subjects taking lipid-lowering drugs before the recruitment are permitted to enter the secondary screening after a 4-week washout period, to allow for sufficient elimination. Eighty-four eligible participants will be randomly assigned to either the FPU treatment group or the sham-treatment group, at a ratio of 2:1.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females aged 18-70 years old.
2. Each side of caudal perirenal fat volume >8000mm3（measured by ultrasound).
3. Low and medium-risk of arteriosclerotic cardiovascular disease (ASCVD) with 3.4 ≤ LDL-C < 4.9 mmol/L or 5.2 ≤ TC < 7.2 mmol/L, as defined by the Chinese guidelines for the management of dyslipidemia in adults(revised edition 2016).
4. Participants should be willing to sign the informed consent form of the study.

Exclusion Criteria:

1. Familial hyperlipidemia.
2. Participants are taking cholesterol metabolism related drugs (e.g. fibrate drugs, thiazide diuretics, glucocorticoid, para-amino salicylic acid, colchicine, thyroid hormone, thyroid preparation, hypoglycemic, heparin, new oral anticoagulant, chlortetracycline, kanamycin, neomycin).
3. Participants are unwilling to stop taking statins.
4. Presence of history of hypertension and at least 2 of the following risk factors:

   * History of smoking (more than 10 years and more than 10 cigarettes per day).
   * Male ≥ 45 years old, female ≥ 55 years old.
   * HDL-C≤1 mmol/L.
5. Presence of clinical documented atherosclerotic cardiovascular diseases (including acute coronary syndrome, stable angina, coronary revascularization, ischemic cardiomyopathy, stroke, transient cerebral ischemia and peripheral atherosclerosis disease defined as stenosis ≥50% or complex plaques of lower limb arteries, renal arteries, carotid arteries and other peripheral arteries).
6. Presence of cardiovascular diseases(e.g. all types of atrial fibrillation; severe structural heart disease including severe pulmonary hypertension resulting from severe aortic or ventricular septal defect, complicated anomaly and severe valvular disease; second degree or above heart block).
7. Presence of previous surgery of kidney or pararenal tissue.
8. Presence of endocrine-related diseases(e.g. Diabetes, Cushing syndrome, thyroidectomy or thyroid dysfunction in need of drug treatment, primary aldosteronism, Hypofunction of adrenal cortex, Polycystic Ovary Syndrome, Hyperparathyroidism, Insulin tumor, Zollinger-Ellison syndrome).
9. Presence of autoimmune diseases (e.g. systemic lupus erythematosus, rheumatoid arthritis, Sjögren syndrome, scleroderma, ulcerative colitis, dermatomyositis, pemphigus, mixed connective tissue disease, sarcoidosis, Takayasu Arteritis).
10. Presence of severe hematologic diseases (e.g. leukemia, lymphoma, aplastic anemia, autoimmune hemolytic anemia, multiple myeloma, Primary Immune Thrombocytopenia, thrombotic thrombocytopenic Purpura, abnormal coagulation).
11. Presence of infectious diseases (e.g. Hepatitis, tuberculosis, AIDS, syphilis, malaria, measles).
12. Presence of parasitic diseases.
13. Presence of significant liver dysfunction (ALT or AST elevation greater than 2 times normal upper limit or other evidence of liver injury).
14. Presence of significant renal dysfunction (GFR< 90 mL / min / 1.73 m2 or other evidence of renal injury).
15. Presence of urinary calculi and/or hematuria (gross hematuria or occult blood positive).
16. Presence of skin infection at the waist.
17. Presence of active malignancy.
18. Pregnant women or in suckling period or planning for pregnancy in trial period.
19. Participants are unwilling to sign an informed consent form.
20. Participants are unable or unwilling to complete follow-up evaluations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The difference in low-density lipoprotein cholesterol (LDL-C) levels between the FPU-treatment and sham treatment groups from baseline to 3 months post-procedure | Day 0 (baseline) to 3-month (end of follow-up)
  The difference in LDL-C levels between the FPU-treatment and sham treatment groups from baseline to 3 months post-procedure.
Incidence of all-cause deaths and serious adverse events | Day 0 (baseline) to 3-month (end of follow-up)
  Serious adverse events including acute liver failure, acute renal failure, acute intestinal perforation, severe embolic events and etc.

SECONDARY OUTCOMES:
The differences between the groups in blood lipid profiles (total cholesterol(TC), triglycerides(TG), and high-density lipoprotein cholesterol(HDL-C)) from baseline to 3 months post-procedure. | Day 0 (baseline) to 3-month (end of follow-up)
  The differences between the groups in blood lipid profiles (total cholesterol(TC), triglycerides(TG), and high-density lipoprotein cholesterol(HDL-C)) from baseline to 3 months post-procedure.
Incidence of other adverse events | Day 0 (baseline) to 3-month (end of follow-up)
  Other adverse events including liver dysfunction, renal dysfunction, etc. at 3 months post-procedure. The following are the safety assessments:
  1. General physical examination and vital signs.
  2. Routine blood and urine tests: C-reactive protein (CRP), ALT, AST, urea nitrogen (BUN), creatinine (Cr), and glycosylated haemoglobin (HbAlc).
  3. Image examinations: electrocardiogram (ECG), renal and renal artery ultrasound, and mid-abdomen routine computed tomography (MAR-CT).
  4. AEs (including ALT or AST ≥ 3 times the upper limit of normal, Cr ≥ 1.5 times the upper limit of normal, and other AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Xiangqing Kong, M.D.&PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- JiangSu Province Hospital / The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No